CLINICAL TRIAL: NCT01013090
Title: Fluid Volume-hypotension Association in Elective Cesarean Section Under Neuraxial Anesthesia
Brief Title: Fluid Volume-hypotension Association in Cesarean Under Neuraxial Anesthesia
Acronym: VOHOCUNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMU-200911-MZ020; NJFY09331M041 (Other Grant/Funding Number: Nanjing Medical University)
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Cesarean Section
Keywords: Epidural anesthesia; Spinal anesthesia; Combined spinal-epidural anesthesia; Fluid therapy; Crystalloid; Colloid
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Epidural crystalloid (Active Comparator): Crystalloid (Ringer's Lactate) is given pre-, co- and post-epidural anesthesia in patients undergoing Cesarean section
  Interventions: Drug: Ringer's Lactate
- Epidural colloid (Active Comparator): Colloid (6% hydroxyethyl starch) is given pre-, co- and post-epidural anesthesia in patients undergoing Cesarean section
  Interventions: Drug: Six percent hydroxyethyl starch
- Spinal crystalloid (Active Comparator): Crystalloid (Ringer's Lactate) is given pre-, co- and post-spinal anesthesia in patients undergoing Cesarean section
  Interventions: Drug: Ringer's Lactate
- Spinal colloid (Active Comparator): Colloid (6% hydroxyethyl starch) is given pre-, co- and post-spinal anesthesia in patients undergoing Cesarean section
  Interventions: Drug: Six percent hydroxyethyl starch
- CSEA crystalloid (Active Comparator): Crystalloid (Ringer's Lactate) is given pre-, co- and post-CSEA anesthesia in patients undergoing Cesarean section
  Interventions: Drug: Ringer's Lactate
- CSEA colloid (Active Comparator): Colloid (6% hydroxyethyl starch) is given pre-, co- and post-CSEA anesthesia in patients undergoing Cesarean section
  Interventions: Drug: Six percent hydroxyethyl starch

INTERVENTIONS:
Drug: Ringer's Lactate — Ringer's Lactate 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 15 ml/kg is given to patients pre-, co- and post-neuraxial blocks
  Other Names: Lactated Ringer's solution
  Arms: CSEA crystalloid; Epidural crystalloid; Spinal crystalloid
Drug: Six percent hydroxyethyl starch — Six percent hydroxyethyl starch 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 15 ml/kg is given to patients pre-, co- and post-neuraxial blocks
  Other Names: HES/HAES
  Arms: CSEA colloid; Epidural colloid; Spinal colloid

SUMMARY:
Hypotension resulted from neuraxial block is a common problem, of which is a special issue in patients undergoing Cesarean section. A large number of studies and clinical guidelines suggest that fluid loading, pre- or co-anesthesia, is a promising manner in preventing hypotension. However, it is still a controversy because the fact of a relatively increased blood volume in parturients. In addition, although it is effective of fluid management, it's precise relationship between fluid (crystalloid or colloid) volume and the proportion of hypotension in Cesarean patients under neuraxial anesthesia is still unknown. The investigators designed this trial to clarify the accurate relationship between fluid volume in an escalated manner and the occurrence of hypotension analyzed with a non-linear regression, and wanted to present the 50% effective volume (EV50) of fluid including crystalloid and colloid in preventing hypotension in patients undergoing Cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* 21-40 yr
* First time of delivery
* ASA status I-II
* No premature
* No genetic and infectious diseases
* Chinese

Exclusion Criteria:

* < 21 yr
* > 40 yr
* Subjects with cardiac and pulmonary disorders
* Dislocation of placenta
* Pregnant hypertension
* Allergy to local anesthetics
* Unwilling to cooperation
* Need intraoperative administration of vascular active agents
* With significant delivery side effects
* With contradictions of neuraxial anesthesia

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Rate of hypotension | Anesthesia begin (0 min) to 120 min after anesthesia

SECONDARY OUTCOMES:
Recurrence of hypotension after ephedrine or phenylephrine | Anesthesia begin (0 min) to 120 min after anesthesia
Consumption of ephedrine and phenylephrine | Anesthesia begin (0 min) to 120 min after anesthesia
Duration of hypotension | Anesthesia begin (0 min) to 120 min after anesthesia
Oxygen saturation during hypotension | Anesthesia begin (0 min) to 120 min after anesthesia
One-min and 5-min Apgar scores | The first and fifth minute after cesarean successful delivery
Low umbilical cord pH (artery < 7.20) | At the time of successful delivery (0 min)

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China